CLINICAL TRIAL: NCT04239794
Title: The Influence of Type of Anesthesia on Postoperative Pain After Laparoscopic Colorectal Cancer Surgery: Multi-center Prospective Randomized Controlled Study
Brief Title: The Influence of Type of Anesthesia on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor (full), Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TIVA-IA-Pain
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Colo-rectal Cancer; Anesthesia
Keywords: Postoperative pain; Opioid consumption; Intraoperative anesthesia
MeSH Terms: conditions — Colonic Neoplasms; Pain, Postoperative | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation anesthesia (Active Comparator): Patients are anesthetized with sevoflurane and remifentanil infusion for maintenance of anesthesia during the surgery
  Interventions: Drug: Sevoflurane
- Total intravenous anesthesia (Experimental): Patients are anesthetized with target-controlled intravenous infusion of propofol and remifentanil infusion for maintenance of anesthesia during the surgery
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — General anesthesia during the laparoscopic colorectal surgery is achieved by using a target-controlled intravenous infusion of propofol.
  Other Names: Propofol 2%
  Arms: Total intravenous anesthesia
Drug: Sevoflurane — General anesthesia during the laparoscopic colorectal surgery is achieved by using an inhalation agent (Sevoflurane).
  Other Names: Sevoflurane inhalant product
  Arms: Inhalation anesthesia

SUMMARY:
The investigators designed a multi-center prospective randomized controlled trial to study the influence of the type of anesthesia on postoperative pain after laparoscopic colorectal cancer surgery. Half of the participants will be anesthetized with propofol and remifentanil, while the other half will be anesthetized with sevoflurane and remifentanil during the surgery. The investigators will measure opioid consumption and pain score in the acute postoperative phase.

DETAILED DESCRIPTION:
Previous studies showed that patients receiving total intravenous anesthesia (TIVA) with propofol are associated with less postoperative pain and less opioid consumption compared with inhalation anesthesia. However, some studies showed conflicting results. In colorectal surgery, there are only retrospective studies that showed the analgesic effect of TIVA and inhalation anesthesia. The investigators designed a multi-center prospective randomized controlled trial and hypothesized that TIVA with propofol would be associated with reduced postoperative opioid consumption and less postoperative pain compared with sevoflurane in laparoscopic colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient scheduled for elective laparoscopic colorectal cancer surgery

Exclusion Criteria:

* Pregnant
* Conversion from laparoscopic to open surgery
* Allergy to anesthetics and analgesics
* Previous abdominal surgery
* Chronic pain
* Chronic analgesic usage

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative 24 h opioid consumption | 24 hours after the surgery
  Cumulative opioid consumption for pain control 24 hours after the surgery

SECONDARY OUTCOMES:
Postoperative 48 h opioid consumption | 48 hours after the surgery
  Cumulative opioid consumption for pain control 48 hours after the surgery
Numerical rating scale (NRS) | 24 and 48 hours after the surgery
  Numerical rating scale (NRS) pain score 24 and 48 hours after the surgery. NRS is an 11-point scale for patient self-reporting of pain; 0-10 where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong SSC, Choi SW, Lee Y, Irwin MG, Cheung CW. The analgesic effects of intraoperative total intravenous anesthesia (TIVA) with propofol versus sevoflurane after colorectal surgery. Medicine (Baltimore). 2018 Aug;97(31):e11615. doi: 10.1097/MD.0000000000011615. PMID 30075537